CLINICAL TRIAL: NCT01578018
Title: Tumor Markers in Lung Cancer: DCAMLK-1LK-1: A Pilot Study
Brief Title: Tumor Markers in Lung Cancer: DCAMLK-1LK-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Principal Investigator, Gary Kinasewitz, Principal Investigator, University of Oklahoma
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 16249
Record Dates: First submitted 2012-04-11; First posted 2012-04-16 (Estimated); Last update posted 2012-08-10 (Estimated); Status verified 2012-08

CONDITIONS: Lung Cancer; Smoking
Keywords: lung cancer; smoking
MeSH Terms: conditions — Lung Neoplasms; Smoking | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lung Cancer (Other): Diagnostic
  Interventions: Other: Measure DCAM levels in blood
- Lung Disease (Other): Diagnostic
  Interventions: Other: DCAM levels in blood

INTERVENTIONS:
Other: Measure DCAM levels in blood — Measure DCAM levels in blood
  Other Names: Lung Cancer
  Arms: Lung Cancer
Other: DCAM levels in blood — DCAM levels in blood
  Other Names: Lung Disease
  Arms: Lung Disease

SUMMARY:
DCAMLK1 is a Ca2+ - ca/modulin (CaM) - dependent protein kinase that is a marker of stem cells in colonic crypts. Mutations within the stem cell population are thought to be responsible for the development of most colorectal carcinomas and studies have shown that DCAMLK1 is highly expressed in these tumors. Since the lung is an embryological development of the foregut, the investigators speculate that DCAMLK1 will also be upregulated in lung cancers.

The aim of this pilot study is to measure DCAMLK1 levels in the blood of patients with suspected malignant and benign lung diseases, and to correlate DCAMKL1 levels with smoking status.

DETAILED DESCRIPTION:
In the investigators' preliminary study DCAMKL1 antigen was detected not only in malignant tissue, but also in BAL fluid from patients with benign lung disease. This suggests that DCAMKL1 expression might be induced by smoking or benign lung diseases. To examine this hypothesis, the investigators will compare DCAMLK1 expression in blood from patients with lung cancer to controls who are current or former smokers with benign lung disease.

Previous work has showed that DCAMLK1 is not detectable in the blood of healthy non smoking individuals. To determine whether smoking and or pulmonary inflammation induce DCAMLK1 expression, the investigators will obtain serum samples from 20 control patients with lung disease who are seen in the Chest Clinic at the Oklahoma City VAMC. Smoking histories will be obtained for all participants and DCAMLK1 levels will be correlated with smoking status.

ELIGIBILITY:
Inclusion Criteria:

* >45 years of age

Exclusion Criteria:

* Unable to provide informed consent

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2011-12; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Tumor Markers in Lung Cancer: | 6 months
  DCAMLK-1LK-1 levels will be measured in the blood of patients with Lung Cancer and compared to that of controls with other lung diseases.

CONTACTS AND LOCATIONS:
Overall Officials: Kellie Jones, MD, Principal Investigator — University of Oklahoma
Locations (1):
- VAMC-OKC, Oklahoma City, Oklahoma, United States